CLINICAL TRIAL: NCT02008955
Title: Determination Of Lysine Requirement in Adults Over 60 Years Using the Indicator Amino Acid Oxidation (IAAO) Method
Brief Title: Lysine Requirement of Elderly Men and Women Over 60 Years of Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Senior Scientist, The Research Institute, Hospital for Sick Children, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0019850580 E
Record Dates: First submitted 2013-12-08; First posted 2013-12-11 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: lysine, elderly, amino acid requirement, diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lysine intake at different levels of intake (Experimental): all subjects will receive all 7 of the lysine test levels, assigned in random order.
  Interventions: Dietary Supplement: Lysine intake provided as a milkshake

INTERVENTIONS:
Dietary Supplement: Lysine intake provided as a milkshake — There are 7 different lysine test levels ranging from 10 to 80 mg of lysine per kilogram body weight per day (10 - 80 mg/kg/d)

SUMMARY:
This study aims to determine the requirement for lysine in men and women over the age of 60 years.

Seven different levels of lysine intake will be tested in each subject in random order. Each level of lysine intake will involve a 3-day maintenance diet, with measures (breath, urine, and blood samples) being collected on the third.

DETAILED DESCRIPTION:
Lysine is an amino acid that is essential in the diet. In our body, lysine makes up protein. It is known that as people get older, over the age of 60, our body goes through many changes such as increase in fat mass and decrease in lean mass such as muscle. This is why we are studying how much of the essential amino acid, lysine, the body needs at this particular age.

The indicator amino acid oxidation (IAAO) method is a minimally invasive method for determining essential amino acid requirements.

As essential amino acids cannot be stored in the body, they are either partitioned into protein synthesis or oxidized if in excess. The premise of the IAAO is that when any essential amino acid is limiting in the body then all other amino acids lose their ability to contribute to protein synthesis and are instead oxidized. The method therefore involves providing graded intakes (from deficient to excess) of the test amino acid, lysine, and then measuring the oxidation of another amino acid, which is called the indicator amino acid. This is done by isotopically labelling the indicator amino acid (13C- phenylalanine) and then measuring the appearance of labelled carbon dioxide (13CO2) in breath with the different intakes of the test amino acid, lysine. The requirement for lysine will be determined by the "breakpoint" - the point at which oxidation of 13C- phenylalanine will plateau.

For the study, participants will first participate in a pre-study assessment in which height, weight, body composition (fat mass and muscle mass) and resting energy expenditure and medical history will be assessed. Also, 5 ml of blood will be collected to test for diabetes and kidney function. The purpose of the pre-assessment is to calculate the participant's dietary requirements for the study, and to assess health status, activity level and dietary patterns.

Participants will then participate in up to 7 different 3-day studies that will be separated by a minimum of 1 week between each 3-day study. The first 2 days are adaptation days and participants will consumed the maintenance diet at home as 4 equal meals. The 3rd day is called a study day and participants will consumed 8 hourly formulas; the first 3 are consumed at home and the remaining 5 are consumed at the Clinical Research Centre at the Hospital for Sick Children. Immediately after the 4th meal, 4 baseline breath and 3 baseline urine samples are collected over the period of an hour. After the 5th meal, rate of carbon dioxide production (VCO2) is measured by indirect calorimetry for a period of 20 minutes. The 5th, 6th, 7th, and 8th meal will contain a small amount of isotope labelled phenylalanine (13C phenylalanine). Two and a half hours after the isotope (13C phenylalanine) is given (between meal 7 and 8) 4 plateau breath and 3 plateau urine samples are collected for a period of an hour. Between the 7th and 8th meal, a 15 ml blood sample will be taken - 10 ml will be used to check for glucose and insulin levels and the remaining 5 ml for amino acid analysis.

Breath samples are used to measure the enrichment of isotopic labelled CO2 (13CO2). Urine samples are used to measure the enrichment of isotopic labelled phenylalanine (13C phenylalanine). Through a series of calculations and applying a two-phase regression analysis, we will be able to determine the requirement for lysine.

ELIGIBILITY:
Inclusion Criteria:

* 60 + years old
* non diabetic
* not obese
* willing to participate in the study and completed the screening procedures (height, weight, fasting blood sample and medical history questionnaire)

Exclusion Criteria:

* obese (BMI greater than 30 kg/m2)
* recent history of weight loss or weight gain
* presence of chronic disease or acute illness that could affect protein and AA metabolism (diabetes, cancer, liver or kidney disease, HIV, acute cold or flu, hypo or hyperthyroidism, rheumatoid arthritis treated with anti-inflammatory medications.
* On medications known to affect protein and amino acid metabolism (steroids)
* Inability to tolerate the diet
* Unwilling to have blood drawn from a venous access, or using a ventilated hood indirect calorimeter for the purposes of the study.
* Significant coffee consumption of more than 2 cups/day
* Significant alcohol consumption of more than one drink/day
* smoking

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
change in oxidation of phenylalanine in response to increasing lysine intake | 8 hours
  F13CO2

SECONDARY OUTCOMES:
phenylalanine oxidations determined from urinary phenylalanine enrichments | 8 hrs
  phenylalanine oxidation (phe OX)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pencharz, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Rafii M, Chapman K, Owens J, Elango R, Campbell WW, Ball RO, Pencharz PB, Courtney-Martin G. Dietary protein requirement of female adults >65 years determined by the indicator amino acid oxidation technique is higher than current recommendations. J Nutr. 2015 Jan;145(1):18-24. doi: 10.3945/jn.114.197517. Epub 2014 Oct 15. PMID 25320185
- [Derived] Rafii M, Paoletti A, He H, Porto B, Szwiega S, Pencharz PB, Ball RO, Kong D, Xu L, Elango R, Courtney-Martin G. Dietary Lysine Requirements of Older Adults Stratified by Age and Sex. J Nutr. 2024 Jul;154(7):2133-2142. doi: 10.1016/j.tjnut.2024.04.034. Epub 2024 May 11. PMID 38735574